CLINICAL TRIAL: NCT02477189
Title: Retrospective Analysis of the Safety and Effectiveness of Using the Silicone Block in Penile Surgery
Status: Completed | Type: Observational
Sponsor: International Medical Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IMD-0115
Record Dates: First submitted 2015-05-15; First posted 2015-06-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Penile Implant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study Group: This was the group that received the penis implant, consented for participation and completed the follow-up questionnaire.
  Interventions: Procedure: Silicone Block

INTERVENTIONS:
Procedure: Silicone Block

SUMMARY:
This is a retrospective evaluation of all subjects who successfully received implantation of the Silicone Block for correction of soft tissue deformities of the penis. In addition, subjects will be sent a questionnaire to complete that will evaluate the subject's ongoing satisfaction with the implant and any adverse events that may not have been reported to the physician.

ELIGIBILITY:
Inclusion Criteria:

* Successful penile implantation with the Silicone Block. Successful implantation is defined as the successful completion of the implantation procedure.

Exclusion Criteria:

* Medical records for the subject are not available for review or tabulation
* Subject did not comply with pre-operative or post-operative instructions.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men age 22 and older who had a penis implant from 2009-2014
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | Up to 4 years, with an average of 2 years
  Number of adverse events that occurred from implantation through the time of the study.

SECONDARY OUTCOMES:
Self-Esteem Score | 7 days pre-surgery to 90 days post-surgery
  Evaluation of a self-esteem score done pre-surgery and post-surgery
Self-confidence score | 7 days pre-surgery to 90 days post-surgery
  Evaluation of a self-confidence score done pre-surgery and post-surgery
Flaccid penile girth | 7 days pre-surgery to 90 days post-surgery
  Measurement of flaccid penile girth done pre-surgery and post-surgery
Quality of Life Questionnaire | 7 days pre-surgery to 90 days post-surgery
  Measurement of issues with penis size from pre-surgery to post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Allen Kamrava, MD, MBA, Beverly Hills, California, United States